CLINICAL TRIAL: NCT05587244
Title: Multicenter, Prospective Post-Market Clinical Follow-Up Study of the G7® Freedom Constrained Vivacit-E® Liners
Brief Title: G7 Freedom Constrained Vivacit-E Liners
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMG2021-36H
Record Dates: First submitted 2022-10-10; First posted 2022-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Osteoarthritis, Hip; Rheumatoid Arthritis; Non-Union Fracture; Trochanteric Fractures; Femoral Neck Fractures; Avascular Necrosis; Dislocation, Hip
MeSH Terms: conditions — Osteoarthritis, Hip; Arthritis, Rheumatoid; Fractures, Ununited; Hip Fractures; Femoral Neck Fractures; Osteonecrosis; Hip Dislocation | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Intervention Model Description: Multicenter, Prospective, Non-controlled, Non-randomized, Consecutive series of patients, two cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Total Hip Arthroplasty Treatment Group (Experimental): This study will enroll (implant) up to 202 hips in total according to the IFU and surgical technique. Of these, up to 135 will be revision hips and up to 67 will be primary hips. This is a dual cohort study (primary and revision); each subject will receive the G7 Acetabular System with the Freedom Constrained Vivacit-E bearing. To minimize potential bias and to maximize our ability to assess inter-site differences, each study site will target up to 27 primary hip arthroplasties and up to 54 revision hip arthroplasties (not exceed 81 implanted hips or 40% of total study population). Each site is encouraged to enroll (implant) both primary and revision subjects.
  Interventions: Device: Total Hip Arthroplasty with G7 Freedom Constrained Vivacit-E Liners

INTERVENTIONS:
Device: Total Hip Arthroplasty with G7 Freedom Constrained Vivacit-E Liners — Primary and/or Revision total hip arthroplasty with the G7 Freedom Constrained Vivacit-E Liners

SUMMARY:
The main objectives of this study are to confirm the long-term safety, performance, and clinical benefits of the G7 Freedom Constrained Vivacit-E Acetabular Liners in primary and revision total hip arthroplasty.

DETAILED DESCRIPTION:
The main objectives of this study are to confirm the long-term safety, performance, and clinical benefits of the G7 Freedom Constrained Vivacit-E Acetabular Liners in primary and revision total hip arthroplasty.

The primary endpoint is defined by the survival of the implant system at 10 years, which is based on removal of the study device and will be determined using the Kaplan-Meier method. The safety of the system will be assessed by monitoring the frequency and incidence of adverse events. Relation of the events to the implant, instrumentation and/or procedure should be specified.

The secondary endpoints are the assessment of performance and clinical benefits by recording patient-reported clinical outcomes measures (PROMs) as well as radiographic outcomes (if available).

The G7 Vivacit-E Freedom Constrained Liner is indicated for use (per IFU) as a component of a total hip prosthesis in primary and revision patients at high risk of dislocation due to a history of prior dislocation, bone loss, joint or soft tissue laxity, neuromuscular disease, or intraoperative instability, and for whom all other options to constrained acetabular components have been considered.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 to 80 years of age, inclusive
* Patient is skeletally mature
* Patient qualifies for unilateral total hip arthroplasty based on physical exam and medical history including at least one of the following:

  * Non-inflammatory degenerative joint disease, including osteoarthritis and avascular necrosis
  * Rheumatoid arthritis
  * High risk for dislocation
  * Undergoing revision hip arthroplasty
  * Correction of functional deformity
  * In need of treatment of non-union, femoral neck fracture, and trochanteric fractures of the proximal femur with head involvement, unmanageable by other techniques
* Patient is willing and able to complete scheduled follow-up evaluations as described in the protocol and Informed Consent
* Patient, or the patient's legally authorized representative, has participated in the Informed Consent process and is willing and able to sign an IRB approved informed consent

Exclusion Criteria:

* Patient is septic, has an active infection or has osteomyelitis at the affected joint
* Patient has significant osteoporosis as defined by treating surgeon
* Patient has metabolic disorder(s) which may impair bone formation
* Patient has osteomalacia
* Patient has distant foci of infections which may spread to the implant site
* Patient has rapid joint destruction, marked bone loss or bone resorption on pre-operative radiographs
* Patient underwent contralateral THA within 3 months of planned index procedure or has a contralateral THA planned within 3 months of the index procedure
* Patient is undergoing simultaneous bilateral THA
* Patient has vascular insufficiency, muscular atrophy at the implant site or neuromuscular disease which might jeopardize the outcome of the surgery.
* In the opinion of the investigator, patient has any concomitant disease which is likely to jeopardize the functioning or success of the implant
* Patient is known to be pregnant
* The patient is in the vulnerable population group, such as

  * a prisoner
  * a known alcohol or drug abuser
  * mentally incompetent or unable to understand what participation in this study entails

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2037-12 (Estimated); Study Completion 2038-12 (Estimated)

PRIMARY OUTCOMES:
Survival of the study device | 10 years
  Survival (whether or not it is still implanted in the subject) determined using Kaplan Meier method.

SECONDARY OUTCOMES:
Incidence of treatment-emergent Adverse Events (safety) | 10 years
  Safety is assessed by monitoring the frequency and incidence of all adverse events, with particular focus on those that may be related to the study device.
Pain and Functional Performance - Modified Harris Hip Score | 10 years
  The Harris Hip Score evaluates hip function, pain, mobility and daily activity impairment after hip replacement surgery.
  The ten items in the Harris hip score consist of answer choices, awarded a number of points. There are four domains evaluated, as follows:
  * Pain - 1 item which scores between 0 and 44;
  * Function - 7 items, scores are between 0 and 47;
  * Deformity - 1 item which scores either 0 or 4;
  * Range of motion - 1 item which scores between 0 and 5.
  The overall score varies between 0 and 100, where scores closer to 0 are suggestive of impaired hip function and scores closer to 100 indicate positive outcome.
  There are four categories of hip function status:
  * <70: poor hip status;
  * 70 - 79: fair hip status;
  * 80 - 89: good hip status;
  * 90 - 100: excellent hip status.
Pain and Functional Performance - Oxford Hip Score | 10 years
  "The Oxford Hip Score is patient-reported outcome instrument which contains 12 questions on activities of daily living that assess function and residual pain in patients undergoing total hip replacement surgery.
  Grading the Oxford Hip Score 0 to 19-May indicate severe hip arthritis... 20 to 29-May indicate moderate to severe hip arthritis... 30 to 39-May indicate mild to moderate hip arthritis... 40 to 48-May indicate satisfactory joint function..." Oxford Hip Score. (n.d.) Segen's Medical Dictionary. (2011). Retrieved August 19 2022 from https://medical-dictionary.thefreedictionary.com/Oxford+Hip+Score
  Each question is scored from 0 to 4 with 4 being the best outcome. This method, when summed, produces overall scores running from 0 to 48 with 48 being the best outcome. The overall score is reached by simply summing the scores received for individual questions. This results in a continuous score ranging from 0 (most severe symptoms) to 48 (least symptoms).
Euroqol Patient Quality of life measured at 2 years follow-up (EQ-5D-5L) | 10 Years
  The EuroQol five dimensions questionnaire (EQ-5D-5L) is a five dimensional self-assessment that is comprised of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. These five dimensions can be used to index a subject's health utility on a scale of 0 to 1, where 0 is death and 1 is perfect health. The scoring rule for EQ-5D permits scores less than 0, implying that some health states may be worse than death. Note: no VAS measures will be obtained if completed by phone interview.
Radiographic Performance evaluating radiolucency at 5 years follow-up | 5 Years
  X-rays will be evaluated for radiolucency lines to show the number of subjects with radiolucency. Radiolucency refers to structures that are less dense and permit the x-ray beam to pass through them. Radiolucent structures appear dark or black in the radiographic image.
Radiographic Performance evaluating osteolysis at 5 years follow-up | 5 Years
  X-rays will be evaluated for osteolysis to show the number of subjects with osteolysis. Osteolysis is a progressive condition where bone tissue is destroyed. In this process, bones lose minerals (mostly calcium), softens, degenerates and become weaker.
Radiographic Performance evaluating atrophy/hypertrophy at 5 years follow-up | 5 Years
  X-rays will be evaluated for muscular atrophy/hypertrophy. An increase in total mass of a muscle is referred to as as hypertrophy, whereas a decrease in total mass of a muscle is referred to as atrophy.
Radiographic Performance evaluating component migration at 5 years follow-up | 5 Years
  X-rays will be evaluated for component migration to show the number of subjects with migration. Component migration refers to the presence of the device component gradually moving anteriorly, posteriorly, superiorly, or inferiorly in relation to original placement.
Radiographic Performance evaluating device fracture at 5 years follow-up | 5 Years
  Radiographs will be evaluated (up to 5 years) for evidence of device fracture.
Radiographic Performance evaluating heterotopic ossification at 5 years follow-up | 5 Years
  X-rays will be evaluated for heterotopic ossification to show the number of subjects with heterotopic ossification. Heterotopic ossification refers to the presence of bone in soft tissue where bone normally does not exist (extraskeletal bone).

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Overholser, Study Director — Zimmer Biomet
Locations (10):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Southern California, Los Angeles, California
  - University of Florida Board of Trustees, Gainesville, Florida
  - Jersey City Medical Center, Inc, Livingston, New Jersey
  - The Ohio State University, Columbus, Ohio
  - TOA Research Foundation, Knoxville, Tennessee
  - The University of Texas Health Science Center of Houston, Houston, Texas
  - Medical City Plano, Plano, Texas
  - University of Utah, Salt Lake City, Utah
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No